CLINICAL TRIAL: NCT02278354
Title: 18F-AV-1451 PET Imaging in Professional Fighters
Brief Title: Tau Imaging in Professional Fighters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A11
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Professional Fighters (Experimental): Active professional fighters (with and without cognitive impairment) receiving a flortaucipir PET scan
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Retired Professional Fighters (Experimental): Retired professional fighters (with and without cognitive impairment) receiving a flortaucipir PET scan
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 370 megabecquerel (MBq) (10 mCi)
  Other Names: [F-18]T807; 18F-AV-1451; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain 75-105 minutes post injection

SUMMARY:
Subjects enrolled in the Professional Fighters Brain Health Study (PFBHS) will receive flortaucipir to explore its use as a biomarker for brain injury related to repetitive head trauma and to examine the relationship between clinical presentation and tau deposition.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Currently enrolled in the PFBHS protocol and have participated in a minimum of 10 professional fights
* Can tolerate Positron Emission Tomography (PET) scan procedures
* Have the ability to provide informed consent

Subjects with cognitive impairment

* Have subjective cognitive complaints or objective decline or impairment as determined by the investigator

Exclusion Criteria:

* Have behavior dysfunction that is likely to interfere with imaging
* Are claustrophobic or otherwise unable to tolerate the imaging procedure
* Have current clinically significant cardiovascular disease or clinically significant abnormalities on screening electrocardiogram
* A history of additional risk factors for Torsades de Pointes (TdP) or are taking drugs that are known to cause QT-prolongation
* Have a current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session
* Have current drug or alcohol dependence or alcohol dependence within the past 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Feb 2015 and Feb 2017
Pre-assignment Details: Five subjects enrolled in the study but did not receive a flortaucipir PET scan (2 active, 3 retired). Two additional subjects in the active fighters group did not have the minimum 10 fights required for inclusion into the study, and therefore were considered not to have completed the study. However, their PET scan results were analyzed.
Period: Overall Study
Arm/Group | Active Professional Fighters | Retired Professional Fighters
Started | 12 | 23
Flortaucipir PET Scan | 10 | 20
Completed | 8 | 20
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — <10 professional fights | 2 | 0

BASELINE CHARACTERISTICS:
Population: Only includes subjects who received a flortaucipir PET scan in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Professional Fighters | Retired Professional Fighters | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.27) | 47.6 (10.21) | 42.3 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 20 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 9 | 10
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 3 | 13 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30
Amyloid status [Count of Participants; unit: Participants] — Amyloid status determined by florbetapir PET scan Population: Per protocol, baseline amyloid status was only obtained for fighters > 50 years of age or with a clinical presentation that suggested a possible Alzheimer's disease diagnosis (n=15)
  Participants
    number analyzed (Participants) | 1 | 14 | 15
    Amyloid negative | 1 | 14 | 15
    Amyloid positive | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir Imaging (Quantitative) Between Cognitive Groups
Description: Standard Uptake Value Ratio (SUVr) by subject enrollment group (cognitive impaired/normal) across weighted cortical average, frontal, temporal, parietal, and occipital brain regions. For SUVr, a value of 1 or lower signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan
Population: Cognitively impaired fighters either had subjective cognitive complaints or objective decline or impairment as determined by the investigator.
Measure: Least Squares Mean (95% Confidence Interval); unit: standardized uptake value ratio (SUVr)
Groups:
- Cognitively Impaired Fighters: Fighters (active and retired) with cognitive impairment at baseline
- Cognitively Normal Fighters: Fighters (active and retired) without cognitive impairment at baseline
Arm/Group | Cognitively Impaired Fighters | Cognitively Normal Fighters
Number analyzed (Participants) | 18 | 12
standardized uptake value ratio (SUVr)
  Weighted cortical average | 1.0048 [0.977 to 1.0327] | 0.971 [0.9401 to 1.002]
  Frontal | 0.9731 [0.9394 to 1.0068] | 0.9357 [0.8983 to 0.9732]
  Temporal | 0.9867 [0.9425 to 1.0309] | 0.9305 [0.8812 to 0.9797]
  Parietal | 0.9472 [0.9097 to 0.9847] | 0.9288 [0.8871 to 0.9705]
  Occipital | 0.9513 [0.912 to 0.9906] | 0.9247 [0.8809 to 0.9684]

2. Primary Outcome: Flortaucipir Imaging (Quantitative) Between Fighter Groups
Description: Standard Uptake Value Ratio (SUVr) by subject enrollment group (active fighter/retired fighter) across weighted cortical average, frontal, temporal, parietal, and occipital brain regions. For SUVr, a value of 1 or lower signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan
Measure: Least Squares Mean (95% Confidence Interval); unit: standardized uptake value ratio (SUVr)
Arm/Group | Active Professional Fighters | Retired Professional Fighters
Number analyzed (Participants) | 10 | 20
standardized uptake value ratio (SUVr)
  Weighted cortical average | 0.9965 [0.963 to 1.0299] | 0.9794 [0.9546 to 1.0042]
  Frontal | 0.9816 [0.9411 to 1.022] | 0.9273 [0.8973 to 0.9572]
  Temporal | 0.9838 [0.9306 to 1.0369] | 0.9334 [0.894 to 0.9728]
  Parietal | 0.9623 [0.9172 to 1.0073] | 0.9137 [0.8803 to 0.9471]
  Occipital | 0.9632 [0.916 to 1.0105] | 0.9127 [0.8777 to 0.9478]

3. Primary Outcome: Flortaucipir Imaging (Qualitative) Between Cognitive Groups
Description: Qualitative read results (no, mild, moderate, or intense uptake) compared between cognitively impaired (CI) and cognitively normal (CN) groups.
Time Frame: baseline scan
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitively Impaired Fighters | Cognitively Normal Fighters
Number analyzed (Participants) | 18 | 12
Participants
  No Uptake | 16 | 12
  Mild Uptake | 2 | 0
  Moderate Uptake | 0 | 0
  Intense Uptake | 0 | 0

4. Primary Outcome: Flortaucipir Imaging (Qualitative) Between Fighter Groups
Description: Qualitative read results (no, mild, moderate, or intense uptake) compared between active and retired fighter groups
Time Frame: baseline scan
Measure: Count of Participants; unit: Participants
Arm/Group | Active Professional Fighters | Retired Professional Fighters
Number analyzed (Participants) | 10 | 20
Participants
  No Uptake | 10 | 18
  Mild Uptake | 0 | 2
  Moderate Uptake | 0 | 0
  Intense Uptake | 0 | 0

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after the last study drug administration.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection. AEs occurring after flortaucipir administration, but outside that window were not recorded in the database, unless considered attributable to flortaucipir injection.
Arm/Group | Active Professional Fighters | Retired Professional Fighters
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Professional Fighters (N=10) | Retired Professional Fighters (N=20)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02278354/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02278354/SAP_001.pdf